CLINICAL TRIAL: NCT04510298
Title: A Pilot, 4-Week, Randomized, Double-Blind, Placebo-Controlled, Inpatient, Multicenter Study of the Safety, Population Pharmacokinetics, and Exploratory Efficacy of SP-624 in Acutely Psychotic Adult Subjects With Schizophrenia
Brief Title: A Study of the Safety, PK, and Exploratory Efficacy of SP-624 in Acutely Psychotic Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtsei Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-624-221
Record Dates: First submitted 2020-07-27; First posted 2020-08-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-624 (Experimental): SP-624 oral capsule, 20 mg once daily
  Interventions: Drug: SP-624
- Placebo (Placebo Comparator): Placebo oral capsule, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-624 — Oral Capsule
  Arms: SP-624
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
This is a Phase 1B clinical study evaluating the safety and exploring the effectiveness of SP-624 as compared to placebo in the treatment of adults with schizophrenia experiencing acute psychosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Is willing and able to provide written informed consent to participate in the study.
* Has an identified reliable informant.
* Is, in the investigator's opinion, suitable for initiating a washout from the subject's current antipsychotic regimen, if applicable, and is willing to abstain from prohibited psychotropic medications in accordance with study requirements.

  * Subjects must meet screening eligibility criteria and be in an inpatient setting prior to discontinuing antipsychotic medications.
  * Subject must be able, in the investigator's opinion, to safely discontinue prohibited psychotropic medications prior to Baseline without increased suicidality.
* Has a primary diagnosis of schizophrenia based on the Diagnostic and Statistical Manual 5th edition (DSM-5) criteria and confirmed by Mini International Neuropsychiatric Interview (MINI) for Psychotic Disorders Studies.
* Is experiencing an acute exacerbation or relapse of symptoms.
* Is in generally good physical health, in the investigator's opinion, based on Screening medical history, physical examination, vital signs, and clinical laboratory values.
* Has a body mass index (BMI) between 18 and 40 kg/m2, inclusive.
* For women of reproductive potential: has a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline.
* For women of reproductive potential and men with female partners of reproductive potential: agrees to remain abstinent from sexual intercourse or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of study drug.

Key Exclusion Criteria:

* Is a woman who is pregnant, breastfeeding, or less than 6 months postpartum at Screening.
* Has any primary DSM-5 disorder other than schizophrenia, as confirmed by the MINI.
* Fails to discontinue prohibited psychotropic medications.
* Has, in the investigator's opinion, a significant risk of violent or destructive behavior.
* Is currently hospitalized involuntarily or incarcerated.
* Has a history or presence of any clinically significant medical condition, disease, or surgical history that could, in the investigator's opinion, jeopardize the safety of the subject or validity of the study data, or interfere with the absorption, distribution, metabolism, or excretion of the study drug.
* Is, in the investigator's opinion, not a suitable candidate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 8 weeks

SECONDARY OUTCOMES:
Number of Participants with Abnormal Clinical Laboratory Values | Up to 4 weeks
  chemistry, hematology, and urinalysis tests will be performed
Change from Baseline in Blood Pressure (mmHg) | Up to 4 weeks
  Blood pressure is measured by sphygmomanometer. Change from baseline measurement will be calculated
Change from Baseline in Pulse Rate (beats per minute) | Up to 4 weeks
  Pulse rate is measured by sphygmomanometer. Change from baseline measurement will be calculated
Change from Baseline in Body Temperature (degrees celsius) | Up to 4 weeks
  Body temperature is measured by oral thermometer. Change from baseline measurement will be calculated
Change from Baseline in Body Weight (kilograms) | Up to 4 weeks
  Body weight is measured by weight scale. Measurement is reported in kilograms. Change from Baseline measurement will be calculated.
Change from Baseline in ECG Heart Rate (beats per minute) | Up to 4 weeks
  Heart rate is measured by 12-lead electrocardiogram (ECG). Change from Baseline measure will be calculated.
Change from Baseline in ECG RR Interval (seconds) | Up to 4 weeks
  RR interval is measured by 12-lead electrocardiogram (ECG). Change from Baseline measurement will be calculated.
Change from Baseline in ECG PR Interval (milliseconds) | Up to 4 weeks
  PR interval is measured by 12-lead electrocardiogram (ECG). Change from Baseline measurement will be calculated.
Change from Baseline in ECG QTcF Interval (milliseconds) | Up to 4 weeks
  QTcF is measured by 12-lead electrocardiogram (ECG). Change from Baseline measurement will be calculated.
Number of Participants with Abnormal Physical Examination Findings | Up to 4 weeks
Number of Participants with treatment-emergent suicidal ideation or behavior | Up to 5 weeks
  Treatment-emergent suicidal ideation and/or behavior will be assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS) assessments
Number of Participants with treatment-emergent abnormal movements | Up to 4 weeks
  Treatment-emergent abnormal movements will be assessed using a battery of movement assessments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research, Garden Grove, California
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No